CLINICAL TRIAL: NCT00497796
Title: A Randomized, Double-blind Study To Assess The Efficacy And Safety Of Prophylactic Use Of Maribavir Versus Oral Ganciclovir For The Prevention Of Cytomegalovirus Disease In Recipients Of Orthotopic Liver Transplants
Brief Title: Maribavir Versus Oral Ganciclovir For The Prevention of Cytomegalovirus (CMV) Disease in Liver Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1263-301; 2007-004729-16 (EudraCT Number); SHP620-301 (Other: Shire)
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus; CMV; prophylaxis; liver; liver transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — maribavir; Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: maribavir
- 2 (Active Comparator)
  Interventions: Drug: ganciclovir

INTERVENTIONS:
Drug: maribavir — 100mg twice a day for 14 weeks.
  Arms: 1
Drug: ganciclovir — 1000mg three times per day for 14 weeks.
  Arms: 2

SUMMARY:
The purpose of this research study is to investigate whether or not oral maribavir is safe and effective compared to oral ganciclovir for preventing CMV disease when administered for up to 14 weeks in patients who have had a liver transplant.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infections remain a significant problem following various types of transplants that are associated with strong immunosuppressive therapy. Maribavir is a new oral anti-CMV drug with a novel mechanism of action compared to currently available anti-CMV drugs. This study will test the safety and efficacy of maribavir for the prevention of CMV disease when given as prophylaxis for up to 14 weeks following orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Orthotopic liver transplant recipient
* Donor CMV seropositive / Recipient CMV seronegative
* Enrolled within 10 days after liver transplant
* Able to swallow tablets

Exclusion Criteria:

* Multiple organ transplant
* HIV infection
* CMV disease
* Use of other anti-CMV therapy at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2009-09-14 (Actual); Study Completion 2009-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (55):
- United States (55):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California at San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic College of Medicine, Jacksonville, Florida
  - Tampa General, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Jewish Hospital Louisville, Louisville, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - NYU School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center- Strong Memorial, Rochester, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Transplant Institute, Memphis, Tennessee
  - Baylor University Medical Center (Dallas), Dallas, Texas
  - Baylor College of Medicine (Houston), Houston, Texas
  - Methodist Hospital, Houston, Texas
  - UT Memorial Hermann Hospital and Texas Liver Center, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Univeristy of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045

RESULTS

PARTICIPANT FLOW:
Groups:
- Maribavir 100 mg BID: Maribavir: 100mg twice a day (BID) for 14 weeks.
- Ganciclovir 1000 mg TID: Ganciclovir: 1000mg three times per (TID) day for 14 weeks.
Period: Overall Study
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Started | 147 | 160
Completed | 62 | 101
Not Completed | 85 | 59
Not completed — Adverse event (not related) | 9 | 9
Not completed — Adverse event (related) | 5 | 4
Not completed — CMV infection or disease treatment | 30 | 4
Not completed — Consent withdrawn | 10 | 3
Not completed — Investigator/sponsor discretion | 31 | 34
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not applicable (randomized not treated) | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Safety (ITT-S) population, defined as all randomized subjects who received at least one dose of study drug, regardless of whether they had any post-baseline evaluations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID | Total
Number analyzed (Participants) | 147 | 156 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9.0) | 53 (8.9) | 54 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 37 | 64
  Male | 120 | 119 | 239
Distribution of age [Count of Participants; unit: Participants]
  18 to 44 years | 19 | 22 | 41
  45 to 64 years | 109 | 123 | 232
  65 to 75 years | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Endpoint Committee (EC)-Confirmed Cytomegalovirus (CMV) Disease Within 6 Months Post-Transplantation
Description: All investigator-determined (protocol-defined) cases of CMV disease (i.e., symptomatic CMV infection or CMV organ disease), were adjudicated by an independent, blinded EC. Symptomatic CMV infection was defined as: CMV infection detected by a positive result from a CMV laboratory assay from at least one central laboratory assay (pp65 antigenemia or CMV DNA polymerase chain reaction [PCR] assay in plasma) and fever >/=38 °C on >/=2 occasions >/=24 hours apart within a 7-day period and at least one of the following: new or increased malaise, two successive measurements of leucopenia (white blood cell [WBC] count <3500/mm3 or a WBC count decrease of 20% if the cell count prior to onset of clinical symptoms was >4000/mm3) >/=24 hours apart, atypical lymphocytosis >/=5%, and thrombocytopenia. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: 6 months post-transplant
Population: The modified Intent-to-Treat (ITT-M) population, defined as all randomized subjects who received at least one dose of study drug and had participated in the study for at least 14 weeks or had the potential to receive 14 weeks of therapy by 12-Feb-2009.
Measure: Number; unit: number of participants with event
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
number of participants with event | 14 | 10
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Test type: Non-Inferiority or Equivalence — Based on the ICH guidance, the hypothesis of non-inferiority can be tested using a one-sided 97.5% confidence interval's (CI) upper bound comparing with the non-inferiority margin of 5% (0.05); Rate difference = 0.041, 95% CI 2-sided [-0.038 to 0.119] — Rate difference is the rate of maribavir minus the rate of ganciclovir
Statistical Analysis 2: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Test type: Superiority or Other; p = 0.2754, Cochran-Mantel-Haenszel — The p-value is from the Cochran-Mantel-Haenszel test, adjusting for receipt of induction ALA and geographic region (US or Europe); Odds Ratio (OR) = 1.586, 95% CI 2-sided [0.682 to 3.690]

2. Secondary Outcome: Number of Participants With CMV Infection or EC-confirmed CMV Disease Within 6 Months Post-Transplantation
Description: Incidence of CMV infection or EC-confirmed CMV disease within the 6-month post-transplant period included in this section were defined (1) with infection assessed by pp65 antigenemia assay; (2) with infection assessed by CMV DNA PCR; (3) with infection assessed by either assay (pp65 antigenemia or CMV DNA PCR); and (4) with infection assessed by initiation of anti-CMV therapy.
Time Frame: 6 months post-transplant
Population: The ITT-M population, defined as all randomized subjects who received at least one dose of study drug and had participated in the study for at least 14 weeks or had the potential to receive 14 weeks of therapy by 12-Feb-2009.
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
participants
  pp65 antigenemia assay | 63 | 49
  CMV DNA PCR assay | 72 | 52
  pp65 antigenemia or CMV DNA PCR assay | 81 | 64
  Initiation of anti-CMV therapy | 46 | 39
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of the pp65 antigenemia assay; Test type: Superiority or Other; p = 0.0283, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.793, 95% CI 2-sided [1.065 to 3.020] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 2: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of CMV DNA PCR assay; Test type: Superiority or Other; p = 0.0024, Cochran-Mantel-Haenszel; The p-value is from the Cochran-Mantel-Haenszel test, adjusting for receipt of induction ALA and geographic region (US or Europe); Odds Ratio (OR) = 2.284, 95% CI 2-sided [1.338 to 3.900] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 3: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of pp65 antigenemia or CMV DNA PCR assay; Test type: Superiority or Other; p = 0.0053, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.177, 95% CI 2-sided [1.259 to 3.767] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 4: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of initiation of anti-CMV therapy; Test type: Superiority or Other; p = 0.2339, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.388, 95% CI 2-sided [0.811 to 2.377] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir

3. Secondary Outcome: Time to Onset of CMV Infection or EC-confirmed CMV Disease Within 6 Months Post-Transplantation
Description: All investigator-determined (protocol-defined) cases of CMV disease (i.e., symptomatic CMV infection or CMV organ disease) were adjudicated by an independent, blinded EC. CMV infection was assessed by pp65 Antigenemia or CMV DNA PCR from a central or local lab. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: 6 months post-transplant
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
days | 45 [41 to 68] | 127 [125 to 161]
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of time to onset; Test type: Superiority or Other; p < 0.0001, Log Rank; Adjusted Hazard Ratio = 2.25, 95% CI 2-sided [1.62 to 3.14] — Maribavir versus ganciclovir; Cox's proportional hazards regression model: time = receipt of induction ALA and geographic region (US or Europe) + treatment

4. Secondary Outcome: Number of Participants With Investigator-determined CMV Disease
Description: Symptomatic CMV infection was defined as: CMV infection detected by a positive result from a CMV laboratory assay from at least one central laboratory assay (pp65 antigenemia or CMV DNA polymerase chain reaction [PCR] assay in plasma) and fever >/=38 °C on >/=2 occasions >/=24 hours apart within a 7-day period and at least one of the following: new or increased malaise, two successive measurements of leucopenia (white blood cell [WBC] count <3500/mm3 or a WBC count decrease of 20% if the cell count prior to onset of clinical symptoms was >4000/mm3) >/=24 hours apart, atypical lymphocytosis >/=5%, and thrombocytopenia. CMV organ disease was defined as described by Ljungman et al., 2002.
Time Frame: Through 6 months post-transplant (Day 1 to 100 days and 6 months post-transplant)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
participants
  100 days post-transplant | 17 | 3
  6 months post-transplant | 22 | 18
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of 100 days post-transplant; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of 6 months post-transplant; Test type: Superiority or Other; p = 0.3742, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Number of Participants With EC-confirmed CMV Disease Within 100 Days Post-Transplantation
Description: as for outcome 1
Time Frame: 100 days post-transplant
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
participants | 10 | 0
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Number of Participants With CMV Infection or EC-confirmed CMV Disease Within 100 Days Post-Transplantation
Description: as for outcome 2
Time Frame: 100 days post-transplant
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 113 | 120
participants
  pp65 antigenemia assay | 49 | 19
  CMV DNA PCR assay | 59 | 18
  pp65 antigenemia or CMV DNA PCR assay | 68 | 24
  Initiation of anti-CMV therapy | 37 | 5
Statistical Analysis 1: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of pp65 antigenemia assay; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.041, 95% CI 2-sided [2.179 to 7.494] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 2: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of CMV DNA PCR assay; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.448, 95% CI 2-sided [3.404 to 12.213] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 3: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of pp65 antigenemia or CMV DNA PCR assay; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.020, 95% CI 2-sided [3.342 to 10.843] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir
Statistical Analysis 4: Comparison: Maribavir 100 mg BID vs Ganciclovir 1000 mg TID; Analysis of initiation of anti-CMV therapy; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 11.165, 95% CI 2-sided [4.146 to 30.069] — Mantel-Haenszel odds ratio for maribavir versus ganciclovir

7. Secondary Outcome: Number of Participants With Retransplantation
Time Frame: Through 6 months post-transplant (From Day 1 to 100 days and 6 months post-transplant)
Population: The ITT-Safety (ITT-S) population, defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 147 | 156
participants
  At 100 days post-transplant | 1 | 2
  At 6 months post-transplant | 2 | 2

8. Secondary Outcome: Number of Participants With Graft Failure Related Death
Time Frame: Through 6 months post-transplant (From Day 1 to 100 days and 6 months post-transplant)
Population: The ITT-S population, defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 147 | 156
participants
  100 days post-transplant | 0 | 2
  6 months post-transplant | 1 | 2

9. Secondary Outcome: Number of Participants With Acute Graft Rejection
Description: Rejection was assessed by examining a liver biopsy sample. Diagnosis of graft rejection included a global assessment grade and a rejection activity index score.
Time Frame: 26 weeks post-transplant
Population: The ITT-S population, defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 147 | 156
participants
  100 days post-transplant | 16 | 19
  6 months post-transplant | 20 | 23

10. Secondary Outcome: Number of Participants Who Died Within 6 Months Post-Transplantation
Time Frame: 6 months post-transplant
Population: The ITT-S population, defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 147 | 156
participants | 9 | 6

11. Secondary Outcome: Percent of Participants With Signs of Bone Marrow Suppression
Description: Bone marrow suppression was assessed by the occurrence of adverse events (AEs) of investigator-reported leukopenia, neutropenia, thrombocytopenia, and pancytopenia; absolute neutrophil count (ANC) <1000/mm3; white blood cell (WBC) count toxicity grade shifts from 0-2 at baseline to a maximum of 3-4 post-baseline; and use of hematopoietic growth factors during the 6 month post-transplant period.
Time Frame: 15 weeks
Population: The ITT-S population, defined as all participants who received at least one dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Number analyzed (Participants) | 147 | 156
percent of participants
  Hematology AEs | 14 | 21
  ANC <1000/mm3 | 9 | 16
  WBC count toxicity grade shifts | 16 | 21
  Use of hematopoietic growth factors | 15 | 20

12. Secondary Outcome: Plasma Concentration of Maribavir During Treatment
Description: For the first 16 subjects to have PK profiling performed, PK sampling was collected at Weeks 2, 6 and 10. For subsequent subjects that have PK profiling performed, PK sampling was collected at Weeks 2 and 6. Samples were collected 12 hours after the morning dose of maribavir. Permissible assessment windows for pharmacokinetic profile sampling purposes were +/- 5 days for each sampling day. Samples for determination of maribavir concentration were analyzed by a validated liquid chromatography tandem mass spectrometry (LC/MS/MS) method. For plasma, the minimum detectable concentration for maribavir was 0.2 μg/mL.
Time Frame: 12 hours post-dose after 2, 6, and 10 weeks of treatment
Population: The Pharmacokinetic (PK) population, defined as those participants in the ITT-S population from whom plasma samples were drawn, tested for maribavir concentrations, and complete, evaluable PK data were available.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Maribavir 100 mg BID
Number analyzed (Participants) | 11
μg/mL
  2 weeks, n=10 | 1.65 (2.01)
  6 weeks, n=7 | 1.36 (1.25)
  10 weeks, n=8 | 1.55 (1.17)

13. Secondary Outcome: Plasma Concentration of Maribavir Metabolite VP 44469 During Treatment
Description: For the first 16 subjects to have PK profiling performed, PK sampling was collected at Weeks 2, 6 and 10. For subsequent subjects that have PK profiling performed, PK sampling was collected at Weeks 2 and 6. Samples were collected 12 hours after the morning dose of maribavir. Permissible assessment windows for pharmacokinetic profile sampling purposes were +/- 5 days for each sampling day. Samples for determination of VP 44469 (a metabolite of maribavir) concentration were analyzed by a validated liquid chromatography tandem mass spectrometry (LC/MS/MS) method. For plasma, the minimum detectable concentration for VP 44469 was 0.2 μg/mL.
Time Frame: 12 hours post-dose after 2, 6, and 10 weeks of treatment
Population: The PK population, defined as those participants in the ITT-S population from whom plasma samples were drawn, tested for maribavir concentrations, and complete, evaluable PK data were available.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Maribavir 100 mg BID
Number analyzed (Participants) | 11
μg/mL
  2 weeks, n=10 | 0.609 (0.648)
  6 weeks, n=7 | 0.506 (0.224)
  10 weeks, n=8 | 0.666 (0.656)

ADVERSE EVENTS:
Arm/Group | Maribavir 100 mg BID | Ganciclovir 1000 mg TID
Serious Adverse Events (participants affected / at risk) | 71/147 | 76/156
Other Adverse Events (participants affected / at risk) | 127/147 | 140/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir 100 mg BID (N=147) | Ganciclovir 1000 mg TID (N=156)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0
Diabetes Mellitus (Endocrine disorders) | 2 | 0
Cataract (Eye disorders) | 1 | 0
Ulcerative Keratitis (Eye disorders) | 1 | 0
Abdominal Abscess (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 1
Clostridium Difficile Colitis (Gastrointestinal disorders) | 3 | 3
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Fungal Peritonitis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 3
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0
Oesophageal Candidiasis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Peritonitis (Gastrointestinal disorders) | 1 | 2
Umbilical Hernia (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 7
Alcoholic Liver Disease (Hepatobiliary disorders) | 1 | 0
Ascites (Hepatobiliary disorders) | 3 | 4
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 4 | 2
Cholangitis (Hepatobiliary disorders) | 3 | 2
Cholestasis (Hepatobiliary disorders) | 3 | 0
Cytolytic Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic Artery Aneurysm (Hepatobiliary disorders) | 0 | 2
Hepatic Artery Occlusion (Hepatobiliary disorders) | 0 | 2
Hepatic Artery Stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 1 | 3
Hepatic Haematoma (Hepatobiliary disorders) | 1 | 0
Hepatic Necrosis (Hepatobiliary disorders) | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis C (Hepatobiliary disorders) | 2 | 3
Liver Abscess (Hepatobiliary disorders) | 1 | 1
Portal Hypertension (Hepatobiliary disorders) | 0 | 1
Post Procedural Bile Leak (Hepatobiliary disorders) | 4 | 2
Acute Graft Versus Host Disease (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Liver Transplant Rejection (Immune system disorders) | 4 | 12
Abdominal Sepsis (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1
Cytomegalovirus Gastroenteritis (Infections and infestations) | 2 | 1
Cytomegalovirus Hepatitis (Infections and infestations) | 2 | 0
Cytomegalovirus Infection (Infections and infestations) | 12 | 2
Pneumonia Cytomegaloviral (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 2
Complications Of Transplanted Liver (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Incision Site Cellulitis (Injury, poisoning and procedural complications) | 0 | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Wound Infection (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound Infection (Injury, poisoning and procedural complications) | 3 | 3
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 1
Band Neutrophil Count Increased (Investigations) | 0 | 1
Biopsy Liver Abnormal (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 8 | 4
International Normalised Ratio Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis Fungal (Musculoskeletal and connective tissue disorders) | 0 | 1
Femoral Neck Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Hypoglycaemic Seizure (Nervous system disorders) | 0 | 1
Adjustment Disorder (Psychiatric disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 2
Mental Status Changes (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 1
Mesangioproliferative Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Nephritis Interstitial (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 4 | 3
Urinary Tract Infection (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Neoplasm Malignant (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pleural Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia Staphylococcal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Syncytial Virus Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial Haemorrhage (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir 100 mg BID (N=147) | Ganciclovir 1000 mg TID (N=156)
Anaemia (Blood and lymphatic system disorders) | 9 | 13
Leukocytosis (Blood and lymphatic system disorders) | 8 | 5
Leukopenia (Blood and lymphatic system disorders) | 12 | 19
Neutropenia (Blood and lymphatic system disorders) | 8 | 10
Abdominal Distension (Gastrointestinal disorders) | 0 | 8
Abdominal Pain (Gastrointestinal disorders) | 12 | 15
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 8
Constipation (Gastrointestinal disorders) | 9 | 11
Diarrhoea (Gastrointestinal disorders) | 41 | 36
Dysgeusia (Gastrointestinal disorders) | 22 | 20
Nausea (Gastrointestinal disorders) | 14 | 28
Vomiting (Gastrointestinal disorders) | 14 | 15
Asthenia (General disorders) | 1 | 8
Fatigue (General disorders) | 10 | 18
Oedema Peripheral (General disorders) | 19 | 15
Pyrexia (General disorders) | 15 | 13
Ascites (Hepatobiliary disorders) | 9 | 7
Bile Duct Stenosis (Hepatobiliary disorders) | 9 | 9
Hepatitis C (Hepatobiliary disorders) | 14 | 7
Liver Transplant Rejection (Immune system disorders) | 11 | 8
Hepatic Enzyme Increased (Investigations) | 16 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 19 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 8
Dizziness (Nervous system disorders) | 3 | 12
Headache (Nervous system disorders) | 20 | 29
Insomnia (Nervous system disorders) | 13 | 17
Tremor (Nervous system disorders) | 25 | 20
Anxiety (Psychiatric disorders) | 11 | 4
Renal Failure (Renal and urinary disorders) | 12 | 11
Urinary Tract Infection (Renal and urinary disorders) | 22 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 12
Rash (Skin and subcutaneous tissue disorders) | 8 | 7
Hypertension (Vascular disorders) | 18 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.